CLINICAL TRIAL: NCT05393037
Title: A Phase 3, Multicenter, Randomized, Double-blind, Active Comparator-Controlled Study to Evaluate the Safety, Tolerability, and Immunogenicity of V116 in Adults Living With HIV
Brief Title: Safety and Immunogenicity of V116 in Adults Living With Human Immunodeficiency Virus (HIV) (V116-007, STRIDE-7)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: V116-007; V116-007 (Other: MSD); 2021-006710-36 (EudraCT Number)
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2025-12

CONDITIONS: Pneumococcal Disease
MeSH Terms: conditions — Pneumococcal Infections | interventions — 23-valent pneumococcal capsular polysaccharide vaccine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- V116 + Placebo (Experimental): Part A: Participants will receive a single intramuscular (IM) dose of V116 on Day 1, and a single IM dose of placebo on Week 8. Part B: Participants will receive a single IM dose of PCV15 between 10 to 18 months after V116.
  Interventions: Biological: V116; Biological: Placebo; Biological: PCV15 - Part B
- PCV15 + PPSV23 (Active Comparator): Participants will receive a single IM dose of PCV15 on Day 1, and a single IM dose of PPSV23 on Week 8.
  Interventions: Biological: PCV15; Biological: PPSV23

INTERVENTIONS:
Biological: V116 — Pneumococcal 21-valent conjugate vaccine with 4 μg of each of the following pneumococcal polysaccharides (PnPs) antigen: 3, 6A, 7F, 8, 9N, 10A, 11A, 12F, 15A, 15C, 16F, 17F, 19A, 20A, 22F, 23A, 23B, 24F, 31, 33F, and 35B in each 0.5 mL sterile solution
  Other Names: Pneumococcal 21-valent Conjugate Vaccine
  Arms: V116 + Placebo
Biological: Placebo — Saline in each 0.5 mL sterile solution
  Arms: V116 + Placebo
Biological: PCV15 — Pneumococcal 15-valent conjugate vaccine with 2 μg of each of the following PnPs antigen: 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; and 4 μg of PnPs antigen 6B in each 0.5 mL sterile suspension
  Other Names: VAXNEUVANCE™;
  Arms: PCV15 + PPSV23
Biological: PPSV23 — Pneumococcal 23-valent polyvalent vaccine with 25 μg of each of the following PnPs antigen: 1, 2, 3, 4, 5, 6B, 7F, 8, 9N, 9V, 10A, 11A, 12F, 14, 15B, 17F, 18C, 19A, 19F, 20, 22F, 23F, and 33F in each 0.5 mL sterile solution
  Other Names: PNEUMOVAX™23
  Arms: PCV15 + PPSV23
Biological: PCV15 - Part B — Pneumococcal 15-valent conjugate vaccine with 2 μg of each of the following PnPs antigen: 1, 3, 4, 5, 6A, 7F, 9V, 14, 18C, 19A, 19F, 22F, 23F, and 33F; and 4 μg of PnPs antigen 6B in each 0.5 mL sterile suspension
  Other Names: VAXNEUVANCE™
  Arms: V116 + Placebo

SUMMARY:
This study will evaluate the safety, tolerability, and immunogenicity of a pneumococcal 21-valent conjugate vaccine (V116) in persons living with human immunodeficiency virus (HIV), for the prevention of pneumococcal disease caused by the serotypes in the vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Is infected with HIV
* Is receiving combination anti-retroviral therapy (ART) for ≥6 weeks before study entry with no intended changes to combination ART therapy for 3 months after randomization.
* Is vaccine-naïve

Exclusion Criteria:

* Has a history of opportunistic infections ≤12 months before the first vaccination
* Has a history of noninfectious acquired immune deficiency syndrome-related illness
* Has a history of active hepatitis
* Has a history of invasive pneumococcal disease (IPD) or other culture-positive pneumococcal disease ≤3 years before Visit 2 (Day 1)
* Has a known hypersensitivity to any component of V116, PCV15, or PPSV23, including diphtheria toxoid
* Has a known or suspected congenital immunodeficiency, functional or anatomic asplenia, or history of autoimmune disease
* Has a coagulation disorder contraindicating intramuscular vaccinations.
* Has a recent illness with fever
* Has a known cancer malignancy that is progressing or has required active treatment <3 years before enrollment
* Had prior administration of PCV15 or PCV20.
* Is expected to receive any pneumococcal vaccine during the study outside of the protocol
* Has received systemic corticosteroids for ≥14 consecutive days and has not completed treatment ≥14 days before receipt of study vaccine
* Is currently receiving immunosuppressive therapy, including chemotherapeutic agents or other immunotherapies/immunomodulators used to treat cancer or other conditions, and interventions associated with organ or bone marrow transplantation, or autoimmune disease
* Has received any non-live vaccine ≤14 days before receipt of any study vaccine or is scheduled to receive any non-live vaccine ≤30 days after receipt of any study vaccine
* Has received any live virus vaccine ≤30 days before receipt of any study vaccine or is scheduled to receive any live virus vaccine ≤30 days after receipt of any study vaccine
* Has received a blood transfusion or blood products, including immunoglobulins ≤6 months before receipt of study vaccine or is scheduled to receive a blood transfusion or blood product ≤30 days after receipt of study vaccine
* Is currently participating in or has participated in an interventional clinical study with an investigational compound or device within 2 months of participating in this current study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 313 (Actual)
Dates: Start 2022-07-13 (Actual); Primary Completion 2023-07-13 (Actual); Study Completion 2024-01-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (20):
- United States (7):
  - Pueblo Family Physicians ( Site 0014), Phoenix, Arizona
  - Whitman-Walker Institute ( Site 0009), Washington D.C., District of Columbia
  - Midway Immunology and Research Center ( Site 0003), Ft. Pierce, Florida
  - Orlando Immunology Center ( Site 0004), Orlando, Florida
  - KC CARE Health Center ( Site 0013), Kansas City, Missouri
  - North Texas Infectious Diseases Consultants, P.A ( Site 0001), Dallas, Texas
  - Texas Center for Infectious Disease Associates ( Site 0011), Fort Worth, Texas
- Belgium (2):
  - CHU Saint-Pierre ( Site 0500), Brussels, Bruxelles-Capitale, Region de
  - Insituut voor tropische Geneeskunde ( Site 0501), Antwerp
- Chile (3):
  - Universidad San Sebastian - Providencia ( Site 0111), Providencia, Region M. de Santiago
  - Universidad de Chile - Hospital Clínico Universidad de Chile ( Site 0107), Santiago, Region M. de Santiago
  - Hospital hernan henriquez aravena de temuco-Unidad de Investigación Clínica ( Site 0101), Temuco, Región de la Araucanía
- France (2):
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0601), Paris
  - Hôpital Saint-Louis ( Site 0600), Paris, Île-de-France Region
- South Africa (4):
  - Josha Research ( Site 0900), Bloemfontein, Free State
  - Perinatal HIV Research Unit (PHRU)-Adult Treatment and Research ( Site 0906), Johannesburg, Gauteng
  - Right To Care Research - Esizayo ( Site 0904), Johannesburg, Gauteng
  - Be Part Yoluntu Centre ( Site 0902), Paarl, Western Cape
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital-Preventive and social ( Site 1100), Bangkok, Bangkok
  - Research Institute for Health Sciences-Research Institute for Health Sciences Building 1 ( Site 1101, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Pathirana J, Ramgopal M, Martin C, Lombaard JJ, Chahin C, Launay O, Ratanasuwan W, Greenberg D, Grijalva CG, Orenstein WA, Shenkerman A, Hall L, Fernsler D, Kim Y, Li J, Platt HL; STRIDE-7 Study Group. Safety, tolerability, and immunogenicity of an adult-specific pneumococcal conjugate vaccine, V116, in people living with HIV (STRIDE-7): a two-part, parallel-group, randomised, active comparator-controlled, international, phase 3 trial. Lancet HIV. 2025 Oct;12(10):e679-e690. doi: 10.1016/S2352-3018(25)00165-1. Epub 2025 Sep 12. PMID 40953572
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://www.trialsummaries.com/Study/StudyDetails?id=26853&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study is conducted in two parts. Part A evaluated V116 and the comparator regimen of PCV15 followed by PPSV23. Part B evaluated PCV15 in participants who received V116 in Part A.
Groups:
- V116 + Placebo (Part A), PCV15 (Part B): Participants received a single intramuscular (IM) dose of V116 on Day 1 and a single IM dose of placebo on Week 8 in Part A. In Part B, a single IM dose of PCV15 was given approximately between 10 to 18 months after V116.
- PCV15 + PPSV23 (Part A): Participants received a single IM dose of PCV15 on Day 1, and a single IM dose of PPSV23 on Week 8 in Part A of the study.
Period: Part A
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Started | 156 | 157
Vaccination 1- V116 | 155 | 0
Vaccination 1- PCV15 | 1 | 156
Vaccination 2- Placebo | 154 | 0
Vaccination 2-PCV15 | 0 | 1
Vaccination 2-PPSV23 | 0 | 151
Completed | 152 | 152
Not Completed | 4 | 5
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 2 | 4
Period: Part B
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Started | 126 | 0
Completed | 125 | 0
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A) | Total
Number analyzed (Participants) | 156 | 157 | 313
Age, Continuous [Mean (Standard Deviation); unit: Years] | 44.0 (12.6) | 46.7 (12.3) | 45.3 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 50 | 92
  Male | 114 | 107 | 221
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 44 | 76
  Not Hispanic or Latino | 124 | 112 | 236
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 21 | 12 | 33
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 62 | 63 | 125
  White | 70 | 79 | 149
  More than one race | 1 | 2 | 3
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Solicited Injection-site AEs From Day 1 Through Day 5 Postvaccination in Part A
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited injection-site AEs after any vaccination was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain.
Time Frame: Up to 5 days after each vaccination in Part A
Population: All participants who were randomized and received at least 1 dose of study intervention. Participants were included in the intervention group according to the study intervention actually received. Two participants received the incorrect study intervention that resulted in a regimen inconsistent with the 2 designated regimens planned in this study. Both participants were excluded from the safety analysis population
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 155 | 155
Percentage of Participants
  Injection site erythema | 3.9 [1.4 to 8.2] | 11.0 [6.5 to 17.0]
  Injection site pain | 50.3 [42.2 to 58.4] | 82.6 [75.7 to 88.2]
  Injection site swelling | 7.1 [3.6 to 12.3] | 20.6 [14.6 to 27.9]

2. Primary Outcome: Percentage of Participants With Solicited Systemic AEs From Day 1 Through Day 5 Postvaccination in Part A
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited systemic AEs was assessed following any vaccination. The solicited systemic AEs assessed were fatigue, headache, myalgia, and pyrexia.
Time Frame: Up to 5 days after each vaccination in Part A
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V116 + Placebo (Part A): Participants received a single intramuscular (IM) dose of V116 on Day 1 and a single IM dose of placebo on Week 8 in part A. In part B, a single IM dose of PCV15 will be given approximately between 10 to 18 months after V116.
Arm/Group | V116 + Placebo (Part A) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 155 | 155
Percentage of Participants
  Fatigue | 30.3 [23.2 to 38.2] | 34.2 [26.8 to 42.2]
  Headache | 21.9 [15.7 to 29.3] | 19.4 [13.5 to 26.5]
  Myalgia | 12.3 [7.5 to 18.5] | 15.5 [10.2 to 22.2]
  Pyrexia | 1.9 [0.4 to 5.6] | 3.2 [1.1 to 7.4]

3. Primary Outcome: Percentage of Participants With Vaccine-related Serious Adverse Events (SAEs) From Day 1 Through the Duration of Participation in Part A
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator. Following any vaccination, the percentage of serious adverse events was assessed.
Time Frame: Up to 194 days in Part A
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V116 + Placebo (Part A), PCV15 (Part B): Participants received a single intramuscular (IM) dose of V116 on Day 1 and a single IM dose of placebo on Week 8 in part A. In part B, a single IM dose of PCV15 will be given approximately between 10 to 18 months after V116.
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 155 | 155
Percentage of Participants | 0.0 [0.0 to 2.4] | 0.0 [0.0 to 2.4]

4. Primary Outcome: Serotype-specific Opsonophagocytic Activity (OPA) Geometric Mean Titers (GMT) Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: Serotype-specific OPA to the 13 serotypes common between V116 and PCV15 + PPSV23 and 8 serotypes unique to V116 were determined using a multiplex opsonophagocytic assay (MOPA). GMT is defined as geometric mean titer (1/dil). Serotype-specific OPA GMTs with 95% confidence intervals are presented.
Time Frame: Up to 114 days
Population: Overall participants analyzed included all randomized participants without protocol deviations that could have substantially impacted the results of the immunogenicity analyses. The number analyzed for each serotype is the subset of overall participants analyzed without protocol deviation such as failure to receive study vaccine, failure to receive correct clinical material as per randomization schedule, or receipt of a prohibited medication or prohibited vaccine prior to study vaccination.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
Titers
  Serotype 3 (Shared): number analyzed (Participants) | 128 | 126
  Serotype 3 (Shared) | 170.7 [132.5 to 220.0] | 172.0 [138.4 to 213.7]
  Serotype 6A (Shared): number analyzed (Participants) | 131 | 123
  Serotype 6A (Shared) | 3896.0 [2929.7 to 5181.1] | 3979.5 [3210.6 to 4932.5]
  Serotype 7F (Shared): number analyzed (Participants) | 135 | 126
  Serotype 7F (Shared) | 3482.3 [2815.8 to 4306.6] | 3275.6 [2658.1 to 4036.6]
  Serotype 8 (Shared): number analyzed (Participants) | 137 | 129
  Serotype 8 (Shared) | 1847.5 [1470.9 to 2320.6] | 2262.9 [1776.5 to 2882.5]
  Serotype 9N (Shared): number analyzed (Participants) | 129 | 126
  Serotype 9N (Shared) | 5763.0 [4552.8 to 7294.7] | 5970.0 [4786.9 to 7445.6]
  Serotype 10A (Shared): number analyzed (Participants) | 137 | 128
  Serotype 10A (Shared) | 3693.0 [2870.2 to 4751.5] | 3652.8 [2731.4 to 4885.1]
  Serotype 11A (Shared): number analyzed (Participants) | 134 | 123
  Serotype 11A (Shared) | 3742.5 [3050.7 to 4591.1] | 1722.3 [1277.1 to 2322.7]
  Serotype 12F (Shared): number analyzed (Participants) | 136 | 128
  Serotype 12F (Shared) | 2585.4 [1993.5 to 3353.0] | 2292.4 [1653.2 to 3178.8]
  Serotype 17F (Shared): number analyzed (Participants) | 135 | 124
  Serotype 17F (Shared) | 8698.6 [7046.1 to 10738.5] | 5886.3 [4489.8 to 7717.1]
  Serotype 19A (Shared): number analyzed (Participants) | 137 | 130
  Serotype 19A (Shared) | 2178.9 [1777.1 to 2671.7] | 2667.0 [2193.2 to 3243.1]
  Serotype 20A (Shared): number analyzed (Participants) | 135 | 130
  Serotype 20A (Shared) | 7249.1 [5854.9 to 8975.4] | 5753.3 [4634.0 to 7143.0]
  Serotype 22F (Shared): number analyzed (Participants) | 129 | 129
  Serotype 22F (Shared) | 3622.4 [2902.8 to 4520.4] | 3979.8 [3214.5 to 4927.1]
  Serotype 33F (Shared): number analyzed (Participants) | 123 | 123
  Serotype 33F (Shared) | 14642.5 [11314.9 to 18948.6] | 11864.5 [9283.8 to 15162.5]
  Serotype 15A (Unique to V116): number analyzed (Participants) | 127 | 124
  Serotype 15A (Unique to V116) | 5859.0 [4684.9 to 7327.4] | 1970.5 [1555.1 to 2496.8]
  Serotype 15C (Unique to V116): number analyzed (Participants) | 131 | 126
  Serotype 15C (Unique to V116) | 5613.0 [4136.7 to 7616.3] | 2438.0 [1791.5 to 3317.7]
  Serotype 16F (Unique to V116): number analyzed (Participants) | 129 | 127
  Serotype 16F (Unique to V116) | 6703.0 [5494.0 to 8178.1] | 1839.0 [1474.3 to 2293.9]
  Serotype 23A (Unique to V116): number analyzed (Participants) | 130 | 111
  Serotype 23A (Unique to V116) | 5053.5 [3781.3 to 6753.5] | 1674.9 [1209.9 to 2318.7]
  Serotype 23B (Unique to V116): number analyzed (Participants) | 135 | 125
  Serotype 23B (Unique to V116) | 1593.8 [1182.7 to 2147.9] | 151.0 [98.1 to 232.6]
  Serotype 24B (Unique to V116): number analyzed (Participants) | 132 | 98
  Serotype 24B (Unique to V116) | 3725.6 [3161.1 to 4391.0] | 567.9 [375.4 to 859.1]
  Serotype 31 (Unique to V116): number analyzed (Participants) | 137 | 125
  Serotype 31 (Unique to V116) | 5699.4 [4435.1 to 7324.2] | 530.8 [364.2 to 773.7]
  Serotype 35B (Unique to V116): number analyzed (Participants) | 135 | 128
  Serotype 35B (Unique to V116) | 11306.2 [9364.7 to 13650.1] | 2977.7 [2425.5 to 3655.8]

5. Secondary Outcome: Serotype-specific Immunoglobulin G (IgG) Geometric Mean Concentration (GMC) Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes common between V116 and PCV15 + PPSV23 and 8 serotypes unique to V116 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay.
Time Frame: Up to 114 days
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: μg/mL
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
μg/mL
  Serotype 3 (Shared): number analyzed (Participants) | 138 | 134
  Serotype 3 (Shared) | 0.50 [0.43 to 0.59] | 0.58 [0.49 to 0.67]
  Serotype 6A (Shared): number analyzed (Participants) | 138 | 133
  Serotype 6A (Shared) | 3.79 [2.77 to 5.18] | 2.80 [2.02 to 3.89]
  Serotype 7F (Shared): number analyzed (Participants) | 138 | 134
  Serotype 7F (Shared) | 2.95 [2.31 to 3.77] | 1.81 [1.49 to 2.21]
  Serotype 8 (Shared): number analyzed (Participants) | 138 | 134
  Serotype 8 (Shared) | 7.05 [5.76 to 8.64] | 8.10 [6.66 to 9.85]
  Serotype 9N (Shared): number analyzed (Participants) | 138 | 134
  Serotype 9N (Shared) | 5.02 [4.01 to 6.28] | 3.36 [2.73 to 4.14]
  Serotype 10A (Shared): number analyzed (Participants) | 138 | 134
  Serotype 10A (Shared) | 7.15 [5.24 to 9.75] | 3.73 [2.78 to 5.00]
  Serotype 11A (Shared): number analyzed (Participants) | 138 | 134
  Serotype 11A (Shared) | 4.40 [3.55 to 5.45] | 2.64 [2.13 to 3.27]
  Serotype 12F (Shared): number analyzed (Participants) | 138 | 134
  Serotype 12F (Shared) | 1.10 [0.83 to 1.47] | 0.71 [0.51 to 0.99]
  Serotype 17F (Shared): number analyzed (Participants) | 138 | 134
  Serotype 17F (Shared) | 10.34 [8.24 to 12.96] | 4.43 [3.49 to 5.61]
  Serotype 19A (Shared): number analyzed (Participants) | 138 | 134
  Serotype 19A (Shared) | 5.96 [4.88 to 7.30] | 5.99 [4.83 to 7.43]
  Serotype 20A (Shared): number analyzed (Participants) | 138 | 134
  Serotype 20A (Shared) | 7.08 [5.60 to 8.95] | 4.94 [3.81 to 6.41]
  Serotype 22F (Shared): number analyzed (Participants) | 138 | 134
  Serotype 22F (Shared) | 3.70 [2.96 to 4.61] | 2.99 [2.40 to 3.72]
  Serotype 33F (Shared): number analyzed (Participants) | 138 | 134
  Serotype 33F (Shared) | 7.55 [5.90 to 9.65] | 5.56 [4.41 to 7.01]
  Serotype 15A (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 15A (Unique to V116) | 5.67 [4.37 to 7.36] | 1.02 [0.80 to 1.31]
  Serotype 15C (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 15C (Unique to V116) | 6.92 [5.15 to 9.29] | 2.68 [2.07 to 3.49]
  Serotype 16F (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 16F (Unique to V116) | 1.55 [1.23 to 1.95] | 0.21 [0.16 to 0.26]
  Serotype 23F (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 23F (Unique to V116) | 2.54 [1.85 to 3.50] | 0.41 [0.30 to 0.55]
  Serotype 23B (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 23B (Unique to V116) | 3.27 [2.51 to 4.25] | 0.99 [0.75 to 1.31]
  Serotype 24F (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 24F (Unique to V116) | 1.80 [1.25 to 2.59] | 0.17 [0.13 to 0.21]
  Serotype 31 (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 31 (Unique to V116) | 2.20 [1.78 to 2.72] | 0.25 [0.20 to 0.31]
  Serotype 35B (Unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 35B (Unique to V116) | 10.26 [7.96 to 13.22] | 0.90 [0.73 to 1.10]

6. Secondary Outcome: Serotype-specific OPA Geometric Mean Fold Rises (GMFRs) Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: Activity for the serotypes contained in V116 and PCV15+PPSV23 (13 serotypes shared with PCV15 and PPSV23 and 8 serotypes unique to V116) was determined using a Multiplexed Opsonophagocytic Assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination with V116 and PCV15 + PPSV23.
Time Frame: Baseline, 30 days post vaccination day 1 (V116), and 30 days post vaccination week 8 (PCV15 + PPSV23)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
Ratio
  Serotype 3 (Shared): number analyzed (Participants) | 121 | 118
  Serotype 3 (Shared) | 5.5 [4.3 to 7.1] | 5.3 [4.3 to 6.7]
  Serotype 6A (Shared): number analyzed (Participants) | 122 | 116
  Serotype 6A (Shared) | 14.3 [10.3 to 19.9] | 15.3 [11.3 to 20.7]
  Serotype 7F (Shared): number analyzed (Participants) | 129 | 120
  Serotype 7F (Shared) | 12.3 [9.1 to 16.3] | 7.4 [5.4 to 10.3]
  Serotype 8 (Shared): number analyzed (Participants) | 136 | 127
  Serotype 8 (Shared) | 11.9 [8.6 to 16.3] | 15.0 [10.4 to 21.8]
  Serotype 9N (Shared): number analyzed (Participants) | 126 | 123
  Serotype 9N (Shared) | 6.7 [5.0 to 8.9] | 5.9 [4.5 to 7.7]
  Serotype 10A (Shared): number analyzed (Participants) | 127 | 114
  Serotype 10A (Shared) | 9.4 [7.1 to 12.6] | 7.4 [5.4 to 10.2]
  Serotype 11A (Shared): number analyzed (Participants) | 125 | 117
  Serotype 11A (Shared) | 9.2 [6.4 to 13.4] | 3.8 [2.7 to 5.3]
  Serotype 12F (Shared): number analyzed (Participants) | 128 | 120
  Serotype 12F (Shared) | 57.3 [42.0 to 78.0] | 46.7 [31.4 to 69.4]
  Serotype 17F (Shared): number analyzed (Participants) | 131 | 119
  Serotype 17F (Shared) | 15.1 [11.2 to 20.2] | 8.5 [6.4 to 11.5]
  Serotype 19A (Shared): number analyzed (Participants) | 132 | 127
  Serotype 19A (Shared) | 5.0 [3.9 to 6.3] | 5.6 [4.4 to 7.2]
  Serotype 20A (Shared): number analyzed (Participants) | 130 | 124
  Serotype 20A (Shared) | 7.1 [5.5 to 9.2] | 4.7 [3.7 to 6.0]
  Serotype 22F(Shared): number analyzed (Participants) | 121 | 113
  Serotype 22F(Shared) | 19.2 [13.2 to 28.1] | 19.3 [12.7 to 29.4]
  Serotype 33F (Shared): number analyzed (Participants) | 113 | 119
  Serotype 33F (Shared) | 7.5 [5.6 to 10.1] | 6.8 [5.2 to 9.1]
  Serotype 15A (Unique to V116): number analyzed (Participants) | 108 | 114
  Serotype 15A (Unique to V116) | 5.7 [4.2 to 7.7] | 1.4 [1.1 to 1.8]
  Serotype 15C (Unique to V116): number analyzed (Participants) | 112 | 107
  Serotype 15C (Unique to V116) | 27.8 [18.7 to 41.4] | 16.3 [10.9 to 24.3]
  Serotype 16F (Unique to V116): number analyzed (Participants) | 125 | 119
  Serotype 16F (Unique to V116) | 6.3 [4.8 to 8.2] | 1.7 [1.4 to 2.0]
  Serotype 23A (Unique to V116): number analyzed (Participants) | 95 | 77
  Serotype 23A (Unique to V116) | 9.0 [6.0 to 13.7] | 2.8 [1.7 to 4.8]
  Serotype 23B (Unique to V116): number analyzed (Participants) | 123 | 118
  Serotype 23B (Unique to V116) | 52.0 [35.7 to 75.6] | 7.2 [4.9 to 10.4]
  Serotype 24F (Unique to V116): number analyzed (Participants) | 91 | 69
  Serotype 24F (Unique to V116) | 5.8 [4.0 to 8.3] | 1.0 [0.8 to 1.3]
  Serotype 31 (Unique to V116): number analyzed (Participants) | 133 | 121
  Serotype 31 (Unique to V116) | 19.9 [13.8 to 28.6] | 1.5 [1.1 to 2.0]
  Serotype 35B (Unique to V116): number analyzed (Participants) | 133 | 125
  Serotype 35B (Unique to V116) | 5.4 [4.3 to 6.8] | 1.3 [1.1 to 1.5]

7. Secondary Outcome: Serotype-specific IgG GMFRs Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes common between V116 and PCV15 + PPSV23 and 8 serotypes unique to V116 were quantitated from participants' sera by a multiplex electrochemiluminescence (ECL) assay. Geometric mean fold rise (GMFR) is the geometric mean of fold rise from baseline to postvaccination with V116 and PCV15 + PPSV23
Time Frame: Baseline, 30 days post vaccination day 1 (V116), and 30 days post vaccination week 8 (PCV15 + PPSV23)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
Ratio
  Serotype 3 (Shared): number analyzed (Participants) | 137 | 133
  Serotype 3 (Shared) | 3.7 [3.2 to 4.3] | 4.0 [3.4 to 4.6]
  Serotype 6A (Shared): number analyzed (Participants) | 137 | 132
  Serotype 6A (Shared) | 11.4 [8.8 to 14.6] | 9.2 [7.1 to 11.8]
  Serotype 7F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 7F (Shared) | 9.1 [7.3 to 11.3] | 5.7 [4.7 to 6.8]
  Serotype 8 (Shared): number analyzed (Participants) | 137 | 133
  Serotype 8 (Shared) | 8.1 [6.5 to 10.1] | 10.0 [7.9 to 12.8]
  Serotype 9N (Shared): number analyzed (Participants) | 137 | 133
  Serotype 9N (Shared) | 10.4 [8.3 to 13.0] | 7.8 [6.3 to 9.6]
  Serotype 10A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 10A (Shared) | 12.2 [9.7 to 15.3] | 8.2 [6.7 to 10.0]
  Serotype 11A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 11A (Shared) | 6.6 [5.5 to 7.9] | 4.5 [3.8 to 5.3]
  Serotype 12F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 12F (Shared) | 9.7 [7.7 to 12.4] | 6.7 [5.1 to 8.8]
  Serotype 17F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 17F (Shared) | 13.8 [11.1 to 17.1] | 7.5 [6.2 to 9.1]
  Serotype 19A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 19A (Shared) | 3.8 [3.2 to 4.6] | 4.8 [4.1 to 5.6]
  Serotype 20A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 20A (Shared) | 7.3 [6.0 to 8.9] | 5.4 [4.5 to 6.5]
  Serotype 22F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 22F (Shared) | 13.7 [10.7 to 17.5] | 10.4 [8.4 to 13.0]
  Serotype 33F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 33F (Shared) | 8.1 [6.6 to 10.0] | 5.9 [4.9 to 7.1]
  Serotype 15A (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 15A (unique to V116) | 16.1 [13.1 to 19.9] | 2.4 [2.1 to 2.8]
  Serotype 15C (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 15C (unique to V116) | 16.6 [13.3 to 20.8] | 6.1 [5.0 to 7.5]
  Serotype 16F (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 16F (unique to V116) | 8.8 [7.3 to 10.7] | 1.4 [1.3 to 1.6]
  Serotype 23A (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 23A (unique to V116) | 15.8 [12.3 to 20.3] | 2.8 [2.3 to 3.4]
  Serotype 23B (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 23B (unique to V116) | 10.0 [8.0 to 12.6] | 3.6 [2.9 to 4.4]
  Serotype 24F (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 24F (unique to V116) | 10.9 [8.3 to 14.2] | 1.0 [0.9 to 1.1]
  Serotype 31 (unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 31 (unique to V116) | 11.6 [9.6 to 14.0] | 1.4 [1.3 to 1.6]
  Serotype 35B (unique to V116): number analyzed (Participants) | 138 | 134
  Serotype 35B (unique to V116) | 11.8 [9.4 to 14.7] | 1.1 [1.0 to 1.1]

8. Secondary Outcome: Percentage of Participants With a >=4-fold Rise in OPA Responses From Baseline (Day 1) to Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: Activity for the serotypes contained in V116 and PCV15+PPSV23 (13 serotypes shared with PCV15 and PPSV23 and 8 serotypes unique to V116) was determined using MOPA. The percentage of participants who had ≥4-fold rise in OPA titers were calculated from baseline to postvaccination with V116 and PCV15 + PPSV23
Time Frame: Baseline, 30 days post vaccination day 1 (V116), and 30 days post vaccination week 8 (PCV15 + PPSV23)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
Percentage of Participants
  Serotype 3 (Shared): number analyzed (Participants) | 121 | 118
  Serotype 3 (Shared) | 58.7 [49.4 to 67.6] | 61.9 [52.5 to 70.6]
  Serotype 6A (Shared): number analyzed (Participants) | 122 | 116
  Serotype 6A (Shared) | 73.8 [65.0 to 81.3] | 80.2 [71.7 to 87.0]
  Serotype 7F (Shared): number analyzed (Participants) | 129 | 120
  Serotype 7F (Shared) | 69.0 [60.3 to 76.8] | 59.2 [49.8 to 68.0]
  Serotype 8 (Shared): number analyzed (Participants) | 136 | 127
  Serotype 8 (Shared) | 66.9 [58.3 to 74.7] | 70.1 [61.3 to 77.9]
  Serotype 9N (Shared): number analyzed (Participants) | 126 | 123
  Serotype 9N (Shared) | 56.3 [47.2 to 65.2] | 57.7 [48.5 to 66.6]
  Serotype 10A (Shared): number analyzed (Participants) | 127 | 114
  Serotype 10A (Shared) | 62.2 [53.2 to 70.7] | 60.5 [50.9 to 69.6]
  Serotype 11A (Shared): number analyzed (Participants) | 125 | 117
  Serotype 11A (Shared) | 53.6 [44.5 to 62.6] | 43.6 [34.4 to 53.1]
  Serotype 12F (Shared): number analyzed (Participants) | 128 | 120
  Serotype 12F (Shared) | 92.2 [86.1 to 96.2] | 83.3 [75.4 to 89.5]
  Serotype 17F (Shared): number analyzed (Participants) | 131 | 119
  Serotype 17F (Shared) | 77.1 [68.9 to 84.0] | 64.7 [55.4 to 73.2]
  Serotype 19A (Shared): number analyzed (Participants) | 132 | 127
  Serotype 19A (Shared) | 49.2 [40.4 to 58.1] | 55.9 [46.8 to 64.7]
  Serotype 20A (Shared): number analyzed (Participants) | 130 | 124
  Serotype 20A (Shared) | 59.2 [50.3 to 67.8] | 49.2 [40.1 to 58.3]
  Serotype 22F (Shared): number analyzed (Participants) | 121 | 113
  Serotype 22F (Shared) | 76.0 [67.4 to 83.3] | 71.7 [62.4 to 79.8]
  Serotype 33F (Shared): number analyzed (Participants) | 113 | 119
  Serotype 33F (Shared) | 61.9 [52.3 to 70.9] | 58.8 [49.4 to 67.8]
  Serotype 15A (Unique to V116): number analyzed (Participants) | 108 | 114
  Serotype 15A (Unique to V116) | 59.3 [49.4 to 68.6] | 21.1 [14.0 to 29.7]
  Serotype 16F (Unique to V116) | 53.6 [44.5 to 62.6] | 16.8 [10.6 to 24.8]
  Serotype 23A (Unique to V116): number analyzed (Participants) | 95 | 77
  Serotype 23A (Unique to V116) | 57.9 [47.3 to 68.0] | 32.5 [22.2 to 44.1]
  Serotype 23B (Unique to V116): number analyzed (Participants) | 123 | 118
  Serotype 23B (Unique to V116) | 87.0 [79.7 to 92.4] | 50.0 [40.7 to 59.3]
  Serotype 24F (Unique to V116): number analyzed (Participants) | 91 | 69
  Serotype 24F (Unique to V116) | 53.8 [43.1 to 64.4] | 7.2 [2.4 to 16.1]
  Serotype 31 (Unique to V116): number analyzed (Participants) | 133 | 121
  Serotype 31 (Unique to V116) | 73.7 [65.3 to 80.9] | 16.5 [10.4 to 24.4]
  Serotype 35B (Unique to V116): number analyzed (Participants) | 133 | 125
  Serotype 35B (Unique to V116) | 55.6 [46.8 to 64.2] | 5.6 [2.3 to 11.2]
  Serotype 15C (Unique to V116): number analyzed (Participants) | 112 | 107
  Serotype 15C (Unique to V116) | 80.4 [71.8 to 87.3] | 71.0 [61.5 to 79.4]

9. Secondary Outcome: Percentage of Participants With a >=4-fold Rise in IgG Responses From Baseline (Day 1) to Postvaccination in Part A for 13 Serotypes Common Between V116 and PCV15 + PPSV23 and 8 Serotypes Unique to V116
Description: The GMC of IgG serotype-specific antibodies to the 13 serotypes common between V116 and PCV15 + PPSV23 and 8 serotypes unique to V116 were quantitated from participants' sera by a multiplex ECL assay. The percentage of participants who had ≥4-fold rise in IgG concentration was calculated from baseline to postvaccination with V116 and PCV15 + PPSV23
Time Frame: Baseline, 30 days post vaccination day 1 (V116), and 30 days post vaccination week 8 (PCV15 + PPSV23)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- PCV15 + PPSV23 (Part A): Participants received a single IM dose of PCV15 on Day 1, and a single IM dose of PPSV23 on Week 8.
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B) | PCV15 + PPSV23 (Part A)
Number analyzed (Participants) | 156 | 156
Percentage of participants
  Serotype 3 (Shared): number analyzed (Participants) | 137 | 133
  Serotype 3 (Shared) | 42.3 [33.9 to 51.1] | 50.4 [41.6 to 59.2]
  Serotype 6A (Shared): number analyzed (Participants) | 137 | 132
  Serotype 6A (Shared) | 70.8 [62.4 to 78.3] | 68.2 [59.5 to 76.0]
  Serotype 7F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 7F (Shared) | 70.1 [61.7 to 77.6] | 57.9 [49.0 to 66.4]
  Serotype 8 (Shared): number analyzed (Participants) | 137 | 133
  Serotype 8 (Shared) | 66.4 [57.9 to 74.3] | 73.7 [65.3 to 80.9]
  Serotype 9N (Shared): number analyzed (Participants) | 137 | 133
  Serotype 9N (Shared) | 75.2 [67.1 to 82.2] | 67.7 [59.0 to 75.5]
  Serotype 10A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 10A (Shared) | 76.6 [68.7 to 83.4] | 68.4 [59.8 to 76.2]
  Serotype 11A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 11A (Shared) | 66.4 [57.9 to 74.3] | 54.1 [45.3 to 62.8]
  Serotype 12F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 12F (Shared) | 67.9 [59.4 to 75.6] | 60.2 [51.3 to 68.5]
  Serotype 17F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 17F (Shared) | 83.9 [76.7 to 89.7] | 73.7 [65.3 to 80.9]
  Serotype 19A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 19A (Shared) | 43.8 [35.3 to 52.5] | 58.6 [49.8 to 67.1]
  Serotype 20A (Shared): number analyzed (Participants) | 137 | 133
  Serotype 20A (Shared) | 67.2 [58.6 to 74.9] | 57.1 [48.3 to 65.7]
  Serotype 22F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 22F (Shared) | 76.6 [68.7 to 83.4] | 78.9 [71.0 to 85.5]
  Serotype 33F (Shared): number analyzed (Participants) | 137 | 133
  Serotype 33F (Shared) | 67.9 [59.4 to 75.6] | 63.2 [54.4 to 71.4]
  Serotype 15A (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 15A (Unique to V116) | 83.9 [76.7 to 89.7] | 21.8 [15.1 to 29.8]
  Serotype 15C (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 15C (Unique to V116) | 82.5 [75.1 to 88.4] | 61.7 [52.8 to 69.9]
  Serotype 16F (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 16F (Unique to V116) | 73.7 [65.5 to 80.9] | 9.0 [4.7 to 15.2]
  Serotype 23A (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 23A (Unique to V116) | 82.5 [75.1 to 88.4] | 29.3 [21.8 to 37.8]
  Serotype 23B (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 23B (Unique to V116) | 72.3 [64.0 to 79.6] | 37.6 [29.3 to 46.4]
  Serotype 24F (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 24F (Unique to V116) | 70.1 [61.7 to 77.6] | 0.0 [0.0 to 2.7]
  Serotype 31 (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 31 (Unique to V116) | 83.2 [75.9 to 89.0] | 6.8 [3.1 to 12.5]
  Serotype 35B (Unique to V116): number analyzed (Participants) | 137 | 133
  Serotype 35B (Unique to V116) | 75.9 [67.9 to 82.8] | 0.8 [0.0 to 4.1]

10. Secondary Outcome: Percentage of Participants With Solicited Injection-site AEs From Day 1 of Part B Through Day 5 Postvaccination in Part B
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited injection-site AEs after any vaccination was assessed. The solicited injection-site AEs assessed were redness/erythema, swelling, and tenderness/pain. Percentage of participants with solicited injection-site AEs from Day 1 of Part B through Day 5 postvaccination in Part B.
Time Frame: Up to 5 days after vaccination in Part B
Population: All participants who were randomized and received at least 1 dose of study intervention in part B. Participants were included in the intervention group according to the study intervention actually received.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Groups:
- V116 + Placebo (Part A), PCV15 (Part B): Participants received a single intramuscular (IM) dose of V116 on Day 1 and a single IM dose of placebo on Week 8 in part A. In part B, a single IM dose of PCV15 was given between 10 to 18 months after V116.
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B)
Number analyzed (Participants) | 126
Percentage of Participants
  Injection site erythema | 3.2 [0.9 to 7.9]
  Injection site pain | 61.9 [52.8 to 70.4]
  Injection site swelling | 6.3 [2.8 to 12.1]

11. Secondary Outcome: Percentage of Participants With Solicited Systemic AEs From Day 1 of Part B Through Day 5 Postvaccination in Part B
Description: An adverse event (AE) is any untoward medical occurrence in a patient or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. The percentage of participants with solicited systemic AEs was assessed following any vaccination. The solicited systemic AEs assessed were fatigue, headache, myalgia, and pyrexia. Percentage of participants with solicited systemic AEs from Day 1 of Part B through Day 5 postvaccination in Part B
Time Frame: Up to 5 days after vaccination in Part B
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B)
Number analyzed (Participants) | 126
Percentage of Participants
  Fatigue | 22.2 [15.3 to 30.5]
  Headache | 14.3 [8.7 to 21.6]
  Myalgia | 11.1 [6.2 to 17.9]
  Pyrexia | 0.8 [0.0 to 4.3]

12. Secondary Outcome: Percentage of Participants With Vaccine-related SAEs From Day 1 of Part B Through the Duration of Participation in Part B
Description: A serious adverse event (SAE) is an AE that is life-threatening, requires or prolongs an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly or birth defect, or is another important medical event deemed such by medical or scientific judgment. Relatedness of an SAE to the study vaccine was determined by the investigator. Following any vaccination, the percentage of serious adverse events was assessed. Percentage of participants with vaccine-related SAEs from Day 1 of Part B through the duration of participation in Part B
Time Frame: Up to 44 days after vaccination in Part B
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | V116 + Placebo (Part A), PCV15 (Part B)
Number analyzed (Participants) | 126
Percentage of Participants | 0.0 [0.0 to 2.9]

ADVERSE EVENTS:
Time Frame: Part A - Non-serious adverse events (NSAEs): Up to 30 days after each vaccination; SAEs and all-cause mortality (ACM): Up to 194 days after the first vaccination Part B - NSAEs: Up to 30 days after vaccination; SAEs and ACM: Up to 44 days after vaccination
Description: The all-cause mortality population includes all randomized participants. The SAE and AE analysis population includes all participants who were randomized and received at least 1 dose of study intervention. Two participants received incorrect study intervention that resulted in a regimen inconsistent with the 2 planned regimens. Both participants were excluded from the safety analysis population.
Groups:
- V116 + Placebo (Part A): Participants received a single intramuscular (IM) dose of V116 on Day 1 and a single IM dose of placebo on Week 8 in Part A.
- V116 + Placebo (Part A), PCV15 (Part B): In Part B, a single IM dose of PCV15 was given approximately between 10 to 18 months after V116 in participant who received V116 in Part A.
Arm/Group | V116 + Placebo (Part A) | PCV15 + PPSV23 (Part A) | V116 + Placebo (Part A), PCV15 (Part B)
All-Cause Mortality (participants affected / at risk) | 1/156 | 0/157 | 0/126
Serious Adverse Events (participants affected / at risk) | 4/155 | 6/155 | 1/126
Other Adverse Events (participants affected / at risk) | 96/155 | 136/155 | 82/126
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 + Placebo (Part A) (N=155) | PCV15 + PPSV23 (Part A) (N=155) | V116 + Placebo (Part A), PCV15 (Part B) (N=126)
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0)
Death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | V116 + Placebo (Part A) (N=155) | PCV15 + PPSV23 (Part A) (N=155) | V116 + Placebo (Part A), PCV15 (Part B) (N=126)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 9 (9) | 0 (0)
Fatigue (General disorders) | 47 (56) | 53 (68) | 28 (28)
Injection site erythema (General disorders) | 6 (8) | 17 (19) | 0 (0)
Injection site pain (General disorders) | 78 (93) | 128 (199) | 78 (78)
Injection site swelling (General disorders) | 11 (13) | 32 (36) | 8 (8)
Myalgia (Musculoskeletal and connective tissue disorders) | 20 (22) | 24 (29) | 14 (14)
Headache (Nervous system disorders) | 38 (48) | 31 (35) | 19 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with ICMJE authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/37/NCT05393037/Prot_SAP_000.pdf